CLINICAL TRIAL: NCT05281861
Title: Evaluation of Marginal Adaptation of Onlay Restorations Constructed From Two Types of Glass Ceramics: A Randomized Clinical Trial
Brief Title: Marginal Evaluation of Zirconia Reinforced Lithium Disilicate Partial Coverage Restoration of Egyptian Posterior Teeth.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Walid Awad Abdelhady, Assistant Lecturer, Department of Crown and Bridge, Al-Azhar University, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V.Ambria Adaptation(679/272)
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Carious Teeth; Adaptation
Keywords: Inlay, Onlay, Partial coverage,
MeSH Terms: conditions — Dental Caries | interventions — lithia disilicate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinded (Patient and outcome assessors)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia reinforced Lithium disilicate (Vita Ambria) ceramic onlay restoration (Experimental): The onlays will be constructed from Zirconia reinforced Lithium disilicate (Vita Ambria) glass ceramic system
  Interventions: Other: Zirconia reinforced Lithium disilicate (Vita Ambria) ceramic onlay restoration
- Lithium disilicate (IPS e-max press) ceramic onlay restoration (Active Comparator): The onlays will be constructed from Lithium disilicate (IPS e-max press) glass ceramic system
  Interventions: Other: Lithium disilicate (IPS e-max press) ceramic onlay restoration

INTERVENTIONS:
Other: Zirconia reinforced Lithium disilicate (Vita Ambria) ceramic onlay restoration — In experimental group, Participants will be restored with onlay ceramic restorations constructed from zirconia reinforced Lithium disilicate (Vita Ambria) glass ceramic
  Arms: Zirconia reinforced Lithium disilicate (Vita Ambria) ceramic onlay restoration
Other: Lithium disilicate (IPS e-max press) ceramic onlay restoration — In control group, Participants will be restored with onlay ceramic restorations constructed from Lithium disilicate (IPS e-max press) glass ceramic
  Arms: Lithium disilicate (IPS e-max press) ceramic onlay restoration

SUMMARY:
Objective: To evaluate the marginal adaptation of the zirconia reinforced lithium disilicate (VITA AMBRIA) glass ceramic Inlay/Onlay compared with lithium disilicate(IPS emax Press) glass ceramic Inlay/Onlay in decayed posterior teeth.

DETAILED DESCRIPTION:
A randomized controlled clinical trial, a double-blind (patient and examiner) is conducted by one trained and calibrated operators who perform all restorative procedures. The restorations will be evaluated by a blind and calibrated two examiner using the FDI (World Dental Federation) criteria. A total of 25 subject will be randomly assigned to each group for a total of 50 subject. The randomization sequence will be generated (www.randomlists.com/team-generator) and to ensure the confidentiality of the allocation, this will be used opaque, sealed and numbered envelopes in series. These will be kept with an independent researcher for the moment of inclusion of the subjects.

Both groups will receive Inlay/Onlay preparation . Digital impression will be taken, wax pattern for the Inlay/Onlay restoration will be designed and milled using CAD/CAM(computer-aided design/computer-aided manufacturing) software. After that, the wax pattern will be invested and final Inlay/Onlay restoration will be constructed from VITA AMBRIA and IPS e.max press ingots according to manufacturing instructions.

ELIGIBILITY:
Inclusion Criteria:

* The patient is healthy.
* 18-50 years old.
* Normal occlusion.
* Good oral hygiene.
* Tooth with complete root apex.
* Tooth with moderate coronal decay.

Exclusion Criteria:

* Patient Incapable of self-care, mental illness, undergoing radiotherapy, diabetic patient, allergy to one of the materials used, pregnancy, smoker, parafunctional habits, poor oral hygiene, severe periodontitis, tooth need vital pulp therapy or surgical crown lengthening or marginal elevation, tooth with enamel or dentin hypoplasia or hypocalcification, Mallaligned or malformed teeth and adjacent or opposing teeth are missed.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Marginal Adaptation | 1 year follow up
  Measuring device: visual and probe.
  According to FDI standard(Grade 1-5), which has been defined as follows:
  Grade 1. Harmonious outline, no gaps, no white or discolored lines. Grade 2. Marginal gap (> 50 μm and < 150 μm), white lines; small marginal fracture removable by polishing; slight ditching, slight step /flashes, minor irregularities Grade 3. Gap (> 150 μm and < 250 μm) not removable; several small marginal fractures; major irregularities, ditching or flash, steps.
  Grade 4. Gap (> 250 μm) dentine/base exposed, chip fracture damaging margins, Notable enamel, or dentine wall fracture.
  Grade 5. Restoration is loose but in situ.

SECONDARY OUTCOMES:
Restoration Fracture and retention | 1 year follow up
  Fracture and retention of the onlay restoration will be evaluated. Measuring device: visual and probe.
  According to FDI standard (Grade 1-5), which has been defined as follows:
  Grade 1: Restoration is present with no fractures, cracks or chipping. Grade 2:Small hairline cracks are visible. Grade 3:Several hairline cracks are present and/or limited chipping of material without damage to marginal quality or proximal contacts.
  Grade 4: Fractures affect marginal quality and/or proximal contacts; bulk fractures with probable gap > 250 μm with or without partial loss of less than half the restoration.
  Grade 5:Loss of restoration or bulk fracture with probable gap > 250 μm with partial loss of the restoration.
Effect of the restoration on the periodontium | 1 year follow up
  inflammation will be evaluated. Measuring device: visual and probe according to
  FDI standard (Grade 1-5), which has been defined as follows:
  Grade 1: No plaque, no inflammation of the gingival papilla. Grade 2: Minimal plaque is present, PBI equivalent to baseline. Grade 3: Difference up to one grade in severity of PBI compared to baseline and in comparison to control tooth.
  Grade 4: Difference of more than one grade of PBI worsening in comparison to control tooth or increase in pocket depth > 1 mm requiring major intervention.
  Grade 5: Severe/ acute gingivitis or periodontitis if related to the restoration requiring immediate replacement of the restoration.
Tooth cracks and fractures | 1 year follow up
  Measuring device: visual and probe according to FDI standard (Grade 1-5) Grade 1: Complete integrity of the restored tooth. Grade 2: Minor marginal crack < 150 μm wide or a hairline crack which cannot be probed. The patient has no clinical symptoms.
  Grade 3:
  (Grade 3.1) Marginal split in the enamel < 250 μm wide. Not possible to remove by polishing without compromising the shape of the tooth surface or damaging the tooth and is left untreated as not expected to cause further damage. (Grade 3.2)Crack < 250 μm. Patient has no or minimal discomfort.
  Grade 4:
  (Grade 4.1) Major marginal split > 250 μm that requires repair and/or dentin or base exposed . (Grade 4.2):A 250-μm probe/explorer can be inserted into a crack Grade 5: A cusp or major tooth fracture requiring immediate replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed FA Metwally, BDS, Study Director — Lecturer of Crown and Bridge Faculty of Dental Medicine, Al-Azhar University; . Khaled MO Haggag, Professor, Study Chair — Professor of Crown and Bridge Faculty of Dental Medicine, Al-Azhar University
Locations (1):
- Al-Azhar University (Cairo), Cairo, Egypt

REFERENCES:
- [Background] Falahchai M, Babaee Hemmati Y, Neshandar Asli H, Neshandar Asli M. Marginal adaptation of zirconia-reinforced lithium silicate overlays with different preparation designs. J Esthet Restor Dent. 2020 Dec;32(8):823-830. doi: 10.1111/jerd.12642. Epub 2020 Aug 18. PMID 32810388
- [Background] Guess PC, Vagkopoulou T, Zhang Y, Wolkewitz M, Strub JR. Marginal and internal fit of heat pressed versus CAD/CAM fabricated all-ceramic onlays after exposure to thermo-mechanical fatigue. J Dent. 2014 Feb;42(2):199-209. doi: 10.1016/j.jdent.2013.10.002. Epub 2013 Oct 24. PMID 24161516
- [Background] Bastos NA, Bitencourt SB, Carneiro RF, Ferrairo BM, Strelhow SSF, Dos Santos DM, Bombonatti JFS. Marginal and internal adaptation of lithium disilicate partial restorations: A systematic review and meta-analysis. J Indian Prosthodont Soc. 2020 Oct-Dec;20(4):338-344. doi: 10.4103/jips.jips_112_20. Epub 2020 Oct 8. PMID 33487960